CLINICAL TRIAL: NCT00167791
Title: Multicenter Trial Using Multi-dose Rituximab as Induction and Desensitization Therapy for Patients on the Waiting List for Kidney Transplant With a Positive Donor Specific Crossmatch to a Living Donor
Brief Title: Rituximab Desensitization Therapy for Patients on the Waiting List for Kidney Transplant
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-2004-0265; RIST
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2014-04

CONDITIONS: End Stage Renal Disease
Keywords: transplant; desensitization; kidney transplant
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: rituximab — Rituximab 375mg/m2 IV weekly times 4 weeks

SUMMARY:
This is a study of patients who have a high risk of kidney rejection before kidney transplant. The hypothesis is that treatment with a medication called rituximab will make it possible for them to receive a kidney transplant from a donor who previously did not present a good match.

ELIGIBILITY:
Inclusion Criteria:

* Active status on a kidney transplant waiting list with positive cross match against a living donor

Exclusion Criteria:

* Receipt of a live vaccine within 4 weeks prior to randomization
* Previous Treatment with Rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Conversion of a positive donor specific cross-match to a living donor to a negative cross-match thereby allowing successful transplantation. | assess 4 weeks after Rituximab treatment completed
Transplant success or failure following the desensitization protocol. | ongoing assessment for 2 years after transplant

SECONDARY OUTCOMES:
Decrease in incidence of humoral rejection to less than 50% at 1 year. | assess 1 year after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda T Becker, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States